CLINICAL TRIAL: NCT01255761
Title: Phase 4, Randomized, 52-Week Study To Evaluate Two Assessment Tools To Predict Treatment Success At 52 Weeks Based On A Treatment Decision At Week 12 In Subjects With Moderate To Severe Rheumatoid Arthritis Receiving Cimzia
Brief Title: A Comparison of Two Assessment Tools in Predicting Treatment Success of Cimzia in Rheumatoid Arthritis Subjects
Acronym: PREDICT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA0064
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab Pegol; Cimzia; Rheumatoid Arthritis; CDAI; RAPID3
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RAPID3 to assess response to Cimzia (Other): RAPID3 is a subject-based assessment tool used to assess subject's response to Cimzia.
  Subjects will be randomized to a patient measure tool, a tool based on patient-report outcomes (RAPID3); using a total score of 30 points
  Interventions: Biological: Certolizumab Pegol (CZP)
- CDAI to assess response to Cimzia (Other): CDAI is an investigator-based assessment tool used to assess subject's response to Cimzia.
  Subjects will be randomized to a clinical measures tool, a tool based on Investigator measures without the need for a lab value (CDAI)
  Interventions: Biological: Certolizumab Pegol (CZP)

INTERVENTIONS:
Biological: Certolizumab Pegol (CZP) — 400 mg subcutaneous injection at Weeks 0, 2 and 4
  200 mg subcutaneous injection every two weeks, Week 6 through Week 52
  Other Names: Cimzia

SUMMARY:
Phase 4 study to evaluate a routine patient completed assessment (RAPID3) compared to a physician completed assessment (CDAI) to predict treatment success with subjects with moderate to severe rheumatoid arthritis

DETAILED DESCRIPTION:
RA0064 is a Phase 4, multicenter, randomized, 52-week study. All eligible subjects will receive open label Cimzia 400 mg at Weeks 0, 2 and 4, followed by Cimzia 200 mg every 2 weeks at Weeks 6 to 50 for the treatment of moderate to severe rheumatoid arthritis. All subjects will be assessed using the 2 assessment tools: the subject-based Routine Assessment of Patient Index (RAPID3) and the investigator-based Clinical Disease Activity Index (CDAI)

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older
* Subjects with a diagnosis of Adult-onset Rheumatoid Arthritis of at least 3 months as defined by the 1987 American College of Rheumatology (ACR) classification criteria
* Subjects with active Rheumatoid Arthritis as defined by:

  * 4 tender joints (28 joint count) at Screening and Baseline Visits; and
  * 4 swollen joints (28 joint count) at Screening and Baseline Visits
* Subjects who have had an unsatisfactory response or intolerance to at least 1 traditional Disease-modifying Antirheumatic Drugs (DMARD)

Exclusion Criteria:

* Subjects must not have a diagnosis of any other inflammatory Arthritis
* Subjects must not have greater than 3 Arthroplasties due to Rheumatoid Arthritis and/or Steinbrocker IV Functional Capacity
* Subjects must not have a secondary non-inflammatory type of Arthritis that would interfere with study evaluation
* Subjects must not be diagnosed with Fibromyalgia with sufficient symptoms requiring treatment
* Subjects must not have a history of Infected Joint Prosthesis
* Subjects must not have discontinued biological therapy for their Rheumatoid Arthritis due to Severe Hypersensitivity Reaction or Anaphylactic Reaction
* Subjects must not have received more than 2 anti- Tumor Necrosis Factor (TNF) agents prior to enrollment
* Subjects must not have received treatment with Abatacept and/or Rituximab or have received any experimental or approved B cell therapeutic agent
* Subjects must not have a history of chronic alcohol or drug abuse
* Subjects must not have known hypersensitivity to any components of the investigational medicinal product
* Subjects must not have a history of chronic infections, recent serious or life-threatening infection within 6 months or any current sign or symptom that may indicate an infection
* Subjects must not have a history of a Blood Dyscrasias
* Subjects with known Tuberculosis (TB) Disease, high risk of acquiring TB or latent TB infection
* Subjects must not be at high risk of infection
* Subjects must not have a history of Lymphoproliferative Disorder including Lymphoma signs and symptoms suggestive of Lymphoproliferative Disease
* Subjects must not have concurrent acute or chronic Viral Hepatitis B or C
* Subjects must not have known Human Immunodeficiency Virus (HIV) infection
* Subject must not have concurrent Malignancy or history of Malignancy
* Subjects must not have a current or recent history of severe, progressive, and/or uncontrolled Renal, Hepatic, Hematological, Gastrointestinal, Endocrine, Pulmonary, Cardiac, Neurological or Cerebral Disease
* Subjects must not have Class III or IV Congestive Heart Failure
* Subjects must not have history of, or suspected Demyelinating Disease of the Central Nervous System
* Subjects must not have a history of adverse reaction to Polyethylene Glycol (PEG)
* Subjects must not have significant laboratory abnormalities which in the investigators judgment would make the subject unsuitable for inclusion
* Subjects must not have a known history or clinically active infection with Histoplasma, Coccidiodes, Paracoccidioides, Pneumocystis, Nontuberculous Mycobacteria, Blastomyces or Aspergillus
* Subject must not have a known history of or be currently diagnosed with Systemic Lupus Erythematosus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (110):
- United States (110):
  - 137, Birmingham, Alabama
  - 166, Huntsville, Alabama
  - 165, Peoria, Arizona
  - 216, Tucson, Arizona
  - 168, Hot Springs, Arkansas
  - 241, Jonesboro, Arkansas
  - 153, Little Rock, Arkansas
  - 111, Covina, California
  - 208, Escondido, California
  - 103, Fullerton, California
  - 155, Huntington Beach, California
  - 202, La Mesa, California
  - 203, Loma Linda, California
  - 233, Los Angeles, California
  - 105, Palm Desert, California
  - 229, Roseville, California
  - 113, Sacramento, California
  - 127, San Diego, California
  - 106, Santa Maria, California
  - 172, Santa Monica, California
  - 212, Upland, California
  - 231, Van Nuys, California
  - 158, Whittier, California
  - 121, Bridgeport, Connecticut
  - 200, Bridgeport, Connecticut
  - 107, Danbury, Connecticut
  - 195, Danbury, Connecticut
  - 138, Hamden, Connecticut
  - 218, Lewes, Delaware
  - 108, Aventura, Florida
  - 120, Dunedin, Florida
  - 101, Ocala, Florida
  - 225, Orange Park, Florida
  - 227, Ormond Beach, Florida
  - 184, Palm Harbor, Florida
  - 145, Sarasota, Florida
  - 191, Tampa, Florida
  - 236, Vero Beach, Florida
  - 144, Atlanta, Georgia
  - 232, Atlanta, Georgia
  - 157, Lawrenceville, Georgia
  - 217, Coeur d'Alene, Idaho
  - 206, Idaho Falls, Idaho
  - 193, Rock Island, Illinois
  - 207, Springfield, Illinois
  - 186, Elizabethtown, Kentucky
  - 204, Lexington, Kentucky
  - 230, Louisville, Kentucky
  - 149, Cumberland, Maryland
  - 237, Hagerstown, Maryland
  - 197, Wheaton, Maryland
  - 118, Mansfield, Massachusetts
  - 132, Worcester, Massachusetts
  - 140, Lansing, Michigan
  - 226, Petoskey, Michigan
  - 114, Saint Clair Shores, Michigan
  - 188, Bridgeton, Missouri
  - 109, St Louis, Missouri
  - 133, St Louis, Missouri
  - 124, Lincoln, Nebraska
  - 205, Reno, Nevada
  - 159, Lebanon, New Hampshire
  - 189, Nashua, New Hampshire
  - 143, Clifton, New Jersey
  - 125, Albuquerque, New Mexico
  - 175, Albany, New York
  - 139, Binghamton, New York
  - 116, Brooklyn, New York
  - 167, Brooklyn, New York
  - 196, Johnson City, New York
  - 174, New York, New York
  - 104, Orchard Park, New York
  - 135, Plainview, New York
  - 215, Rochester, New York
  - 178, Charlotte, North Carolina
  - 210, Durham, North Carolina
  - 234, Hickory, North Carolina
  - 102, Monroe, North Carolina
  - 152, Bethlehem, Pennsylvania
  - 112, Duncansville, Pennsylvania
  - 219, Erie, Pennsylvania
  - 128, Philadelphia, Pennsylvania
  - 147, Sellersville, Pennsylvania
  - 213, Willow Grove, Pennsylvania
  - 235, Wyomissing, Pennsylvania
  - 198, Charleston, South Carolina
  - 228, Columbia, South Carolina
  - 130, Hendersonville, Tennessee
  - 129, Jackson, Tennessee
  - 162, Amarillo, Texas
  - 110, Austin, Texas
  - 156, Austin, Texas
  - 192, Dallas, Texas
  - 185, El Paso, Texas
  - 122, Houston, Texas
  - 170, Houston, Texas
  - 123, Mesquite, Texas
  - 115, Nassau Bay, Texas
  - 117, San Antonio, Texas
  - 119, San Antonio, Texas
  - 161, San Antonio, Texas
  - 190, Victoria, Texas
  - 142, Waco, Texas
  - 136, Burlington, Vermont
  - 146, Arlington, Virginia
  - 150, Chesapeake, Virginia
  - 223, Kennewick, Washington
  - 134, Spokane, Washington
  - 221, Clarksburg, West Virginia
  - 194, Glendale, Wisconsin

REFERENCES:
- [Result] Curtis JR, Herrem C, Ndlovu 'N, O'Brien C, Yazici Y. A somatization comorbidity phenotype impacts response to therapy in rheumatoid arthritis: post-hoc results from the certolizumab pegol phase 4 PREDICT trial. Arthritis Res Ther. 2017 Sep 29;19(1):215. doi: 10.1186/s13075-017-1412-z. PMID 28962590
- [Derived] Curtis JR, Churchill M, Kivitz A, Samad A, Gauer L, Gervitz L, Koetse W, Melin J, Yazici Y. A Randomized Trial Comparing Disease Activity Measures for the Assessment and Prediction of Response in Rheumatoid Arthritis Patients Initiating Certolizumab Pegol. Arthritis Rheumatol. 2015 Dec;67(12):3104-12. doi: 10.1002/art.39322. PMID 26316013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in November 2010. Overall study completion occurred in December 2012.
  The Participant Flow consists of the Randomized Set (RS). The RS consists of all subjects randomized into the study.
  The Baseline Characteristics consists of the Safety Set (SS). SS consists of all subjects that received at least 1 dose of study medication.
Pre-assignment Details: The Full Analysis Set (FAS) consists of all randomized subjects who had a valid Baseline and valid Post-Baseline efficacy measurement.
  FAS-NRI: For all binary efficacy endpoints assessing response, subjects who withdrew early or had a missing assessment were considered nonresponders at that visit. This is known as nonresponse imputation (NRI).
Period: Overall Study
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Started | 369 | 367
Completed | 187 | 192
Not Completed | 182 | 175
Not completed — Adverse Event | 29 | 43
Not completed — Lack of Efficacy | 86 | 74
Not completed — Protocol Violation | 9 | 5
Not completed — Lost to Follow-up | 10 | 8
Not completed — Withdrawal by Subject | 11 | 27
Not completed — Other Reasons | 37 | 18

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics consists of the Safety Set (SS). SS consists of all subjects that received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia | Total
Number analyzed (Participants) | 369 | 367 | 736
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 295 | 276 | 571
  >=65 years | 74 | 90 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.5) | 55.7 (12.8) | 54.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 293 | 573
  Male | 89 | 74 | 163
Region of Enrollment [Number; unit: participants]
  United States | 369 | 367 | 736
Weight [Mean (Standard Deviation); unit: Kilogram] | 84.08 (21.35) | 80.17 (19.23) | 82.13 (20.40)
Height [Mean (Standard Deviation); unit: Centimeters] | 164.94 (9.91) | 164.00 (9.25) | 164.47 (9.59)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/ m^2] | 30.87 (7.23) | 29.82 (6.90) | 30.34 (7.08)

OUTCOME MEASURES:

1. Primary Outcome: Response at Week 12 as Assessed by Randomized Tool [Clinical Disease Activity Index (CDAI) or Routine Assessment of Patient Index Data 3 (RAPID3)]
Description: For subjects randomized to CDAI, response is defined as CDAI ≤10 or 20% improvement from Baseline. For subjects randomized to RAPID3, response is defined as RAPID3 ≤6 or 20% improvement from Baseline.
  CDAI is the sum of tender joint count, swollen joint count, Patient's Global Assessment of Disease Activity as assessed by Multi-dimensional Health Assessment Questionnaire (MDHAQ) subscore, and Investigator's Global Assessment of Disease Activity - VAS (VAS in cm). 28 joints are examined.
  RAPID3 is the sum of the MDHAQ subscores of physical function, pain, and patient's global status.
Time Frame: Baseline (Week 0) to Week 12
Population: Full Analysis Set (FAS) consists of all randomized subjects who had a valid Baseline & valid Post-Baseline efficacy measurement. For all binary efficacy endpoints assessing response, subjects who withdrew early or had a missing assessment at the given visit were considered nonresponders at that visit. This is known as nonresponse imputation (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of participants
  Yes | 64.7 | 76.4
  No | 35.3 | 23.6
Statistical Analysis 1: Comparison: RAPID3 to Assess Response to Cimzia vs CDAI to Assess Response to Cimzia; The null hypothesis was: (Proportion of Rapid 3 responders)-(Proportion of CDAI responders) ≤ delta with a delta of -10 %. A 2-sided 95 % Confidence Interval (CI) for the difference in proportion of responders was computed; Test type: Non-Inferiority or Equivalence — If the lower bound of the 2-sided 95 % CI was greater than -10 %, the null hypothesis was rejected and RAPID3 was deemed comparable to CDAI in assessing response to Certolizumab Pegol therapy at 12 weeks; ANCOVA — Study was intended to show the comparability of RAPID3 with CDAI. Assessment of whether the study objective was met was based on CIs rather than p-values. Both variables need to be significant to claim comparability between the two assessment tools; Difference in proportions from ANCOVA with tool as factor & Baseline DAS28(ESR), gender, age, prior anti-TNF use & disease duration as covariates; Difference in proportion = -0.119, 95% CI 2-sided [-0.184 to -0.053]

2. Primary Outcome: Responders at Week 12 (as Assessed by Randomized Tool Clinical Disease Activity Index [CDAI] or Routine Assessment of Patient Index Data [RAPID3]) Achieving Low Disease Activity (Disease Activity Score 28 [Erythrocyte Sedimentation Rate]≤3.2) at Week 52
Description: For subjects randomized to CDAI, response is defined as CDAI ≤10 or 20% improvement from Baseline. For subjects randomized to RAPID3, response is defined as RAPID3 ≤6 or 20% improvement from Baseline.
  DAS28(ESR) is calculated from the tender joint count, swollen joint count, erythrocyte sedimentation rate (ESR in mm/hour), and Patient's Global Assessment of Disease Activity as assessed by Multi-dimensional Health Assessment Questionnaire (MDHAQ) subscore using this formula: 0.56x√(TJC) + 0.28x√(SJC) + 0.70xlognat (ESR) + 0.014xGlobal Assessment of Arthritis where 28 joints are examined.
Time Frame: Baseline (Week 0) to Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 238 | 279
percentage of participants
  Yes | 31.5 | 32.3
  No | 68.5 | 67.7
Statistical Analysis 1: Comparison: RAPID3 to Assess Response to Cimzia vs CDAI to Assess Response to Cimzia; The null hypothesis was: (Proportion of Rapid 3 responders)-(Proportion of CDAI responders) ≤ delta with a delta of -15 %. A 2-sided 95 % Confidence Interval (CI) for the difference in proportion of responders was computed; Test type: Non-Inferiority or Equivalence — If the lower bound of the 2-sided 95 % CI was greater than -15 %, the null hypothesis was rejected and RAPID3 was deemed comparable to CDAI in assessing percent of Week 12 responders achieving LDA at Week 52; ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in proportion = -0.013, 95% CI 2-sided [-0.093 to 0.066]

3. Secondary Outcome: Percentage of All Subjects Who Are Both Responders at Week 12 and With Non-low Disease Activity (Disease Activity Score 28 [Erythrocyte Sedimentation Rate] > 3.2) at Week 52
Description: as for outcome 2
Time Frame: Baseline (Week 0) to Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of participants
  Yes | 44.3 | 51.8
  No | 55.7 | 48.2

4. Secondary Outcome: Responders at Week 12 Achieving Remission (Disease Activity Score 28 [Erythrocyte Sedimentation Rate] < 2.6) at Week 52
Description: as for outcome 2
Time Frame: Baseline (Week 0) to Week 52
Population: The measurement only includes subjects that were responders at Week 12, and this is the denominator for the percentages.
  The Full Analysis Set (FAS)-Nonresponse imputation (NRI) population set was used for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 238 | 279
percentage of participants
  Yes | 21.8 | 23.3
  No | 78.2 | 76.7

5. Secondary Outcome: Percentage of All Subjects Who Are Both Responders at Week 12 and With Non-remission (Disease Activity Score 28 [Erythrocyte Sedimentation Rate] > 2.6) at Week 52
Description: as for outcome 2
Time Frame: Baseline (Week 0) to Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of participants
  Yes | 50.5 | 58.6
  No | 49.5 | 41.4

6. Secondary Outcome: Change From Baseline in the Disease Activity Score 28 Erythrocyte Sedimentation Rate [DAS28 (ESR)] Assessed at Week 12
Description: The DAS28(ESR) score is a measure of the subject's disease activity.
  DAS28(ESR) is calculated from the tender joint count (28 joints), swollen joint count (28 joints), erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity as assessed by Multi-dimensional Health Assessment Questionnaire (MDHAQ) subscore using this formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined. Lower scores indicate less disease activity.
Time Frame: Baseline (Week 0) to Week 12
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who had a valid Baseline and valid Post-Baseline efficacy measurement. The Last Observation Carried Forward (LOCF) was used for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 355 | 355
units on a scale | -2.20 (1.33) | -2.11 (1.39)

7. Secondary Outcome: Change From Baseline in Disease Activity Score 28 Erythrocyte Sedimentation Rate [DAS28 (ESR)] Assessed at Week 52
Description: as for outcome 6
Time Frame: Baseline (Week 0) to Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 355 | 355
units on a scale | -2.26 (1.45) | -2.14 (1.50)

8. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Assessed at Week 12
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity as assessed by Multi-dimensional Health Assessment Questionnaire (MDHAQ) subscore, and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined.
  The range for the CDAI is 0 - 76 with a negative change in CDAI score indicating an improvement in disease activity and a positive change in score indicating a worsening of disease activity.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 361 | 357
units on a scale | -23.79 (14.35) | -23.11 (14.57)

9. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Assessed at Week 52
Description: as for outcome 8
Time Frame: Baseline (Week 0) to Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 361 | 357
units on a scale | -24.55 (15.42) | -23.16 (15.20)

10. Secondary Outcome: Change From Baseline in Routine Assessment of Patient Index Data 3 (RAPID3) Assessed at Week 12
Description: RAPID3 is the sum of the Multi-dimensional Health Assessment Questionnaire (MDHAQ) subscores of physical function, pain, and patient's global status.
  The range for the RAPID3 is 0 - 30 with a negative change in RAPID3 score indicating an improvement in disease activity and a positive change in score indicating a worsening of disease activity.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 361 | 357
units on a scale | -6.78 (5.94) | -6.47 (6.69)

11. Secondary Outcome: Change From Baseline in Routine Assessment of Patient Index Data 3 (RAPID3) Assessed at Week 52
Description: as for outcome 10
Time Frame: Baseline (Week 0) to Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 361 | 357
units on a scale | -6.36 (6.48) | -6.65 (6.99)

12. Secondary Outcome: Percentage of Subjects With DAS28(ESR) (Disease Activity Score 28 [Erythrocyte Sedimentation Rate]) Low Disease Activity (DAS28[ESR] ≤ 3.2) at Week 12
Description: DAS28(ESR) is calculated from the tender joint count, swollen joint count, erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity as assessed by Multi-dimensional Health Assessment Questionnaire (MDHAQ) subscore, using this formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined. Lower scores indicate less disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 25.0 | 28.2
  No | 75.0 | 71.8

13. Secondary Outcome: Percentage of Subjects With DAS28(ESR) (Disease Activity Score 28 [Erythrocyte Sedimentation Rate]) Low Disease Activity (DAS28[ESR] ≤ 3.2) at Week 52
Description: as for outcome 12
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 21.5 | 24.9
  No | 78.5 | 75.1

14. Secondary Outcome: Percentage of Subjects With DAS28(ESR) (Disease Activity Score 28 [Erythrocyte Sedimentation Rate]) Remission (DAS [ESR] < 2.6) at Week 12
Description: DAS28(ESR) is calculated from the tender joint count, swollen joint count, erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity as assessed by Multi-dimensional Health Assessment Questionnaire (MDHAQ) subscore using this formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined. Lower scores indicate less disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 12.8 | 15.6
  No | 87.2 | 84.4

15. Secondary Outcome: Percentage of Subjects With DAS28(ESR) (Disease Activity Score 28 [Erythrocyte Sedimentation Rate]) Remission (DAS28[ESR] < 2.6) at Week 52
Description: as for outcome 14
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 14.9 | 17.8
  No | 85.1 | 82.2

16. Secondary Outcome: Percentage of Subjects With CDAI (Clinical Disease Activity Index) Low Disease Activity (CDAI ≤ 10) at Week 12
Description: as for outcome 8
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 34.8 | 38.1
  No | 65.2 | 61.9

17. Secondary Outcome: Percentage of Subjects With CDAI (Clinical Disease Activity Index) Low Disease Activity (CDAI ≤ 10) at Week 52
Description: as for outcome 8
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 30.2 | 33.4
  No | 69.8 | 66.6

18. Secondary Outcome: Percentage of Subjects With CDAI (Clinical Disease Activity Index) Remission (CDAI ≤ 2.8) at Week 12
Description: as for outcome 8
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 10.1 | 10.1
  No | 89.9 | 89.9

19. Secondary Outcome: Percentage of Subjects With CDAI (Clinical Disease Activity Index) Remission (CDAI ≤ 2.8) at Week 52
Description: as for outcome 8
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 12.2 | 15.6
  No | 87.8 | 84.4

20. Secondary Outcome: Percentage of Subjects With RAPID3 (Routine Assessment of Patient Index Data) Low Disease Activity (RAPID3 ≤ 6.0) at Week 12
Description: as for outcome 10
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 33.7 | 33.4
  No | 66.3 | 66.6

21. Secondary Outcome: Percentage of Subjects With RAPID3 (Routine Assessment of Patient Index Data) Low Disease Activity (RAPID3 ≤ 6.0) at Week 52
Description: as for outcome 10
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 27.7 | 28.8
  No | 72.3 | 71.2

22. Secondary Outcome: Percentage of Subjects With RAPID3 (Routine Assessment of Patient Index Data) Remission (RAPID3 ≤ 3.0) at Week 12
Description: as for outcome 10
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 14.9 | 18.9
  No | 85.1 | 81.1

23. Secondary Outcome: Percentage of Subjects With RAPID3 (Routine Assessment of Patient Index Data) Remission (RAPID3 ≤ 3.0) at Week 52
Description: as for outcome 10
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 368 | 365
percentage of subjects
  Yes | 18.8 | 20.8
  No | 81.3 | 79.2

24. Secondary Outcome: Number of Work Days Missed (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 12
Description: Number of work days missed in the last month The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 12
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who had a valid Baseline and valid Post-Baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Number of work days missed in last month
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 149 | 134
Number of work days missed in last month | 0.7 (3.6) | 0.7 (3.1)

25. Secondary Outcome: Number of Work Days With Reduced Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 12
Description: Number of work days with reduced productivity in the last month The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Work days with reduced work productivity
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 149 | 134
Work days with reduced work productivity | 1.1 (3.5) | 1.2 (3.5)

26. Secondary Outcome: Interference With Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 12
Description: The arthritis interference in the last month with work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference) The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 149 | 134
units on a scale | 1.7 (2.3) | 1.6 (2.5)

27. Secondary Outcome: Number of Days With No Household Work (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 12
Description: Number of days with no household work in the last month The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days with no household work
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 321 | 314
Days with no household work | 3.2 (5.9) | 3.1 (5.8)

28. Secondary Outcome: Number of Days With Reduced Household Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 12
Description: Number of days with reduced household work productivity in the last month The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days with reduced household work
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 320 | 312
Days with reduced household work | 3.1 (5.7) | 3.1 (5.6)

29. Secondary Outcome: Number of Days Missed of Family/Social/Leisure Activities (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 12
Description: Number of days missed of family/social/leisure activities in the last month The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Activity days missed
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 321 | 314
Activity days missed | 0.7 (2.4) | 0.9 (3.5)

30. Secondary Outcome: Number of Days With Hired Outside Help (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 12
Description: Number of days with hired outside help in the last month The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days with hired outside help
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 321 | 314
Days with hired outside help | 0.4 (2.2) | 0.5 (2.5)

31. Secondary Outcome: Interference With Household Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 12
Description: The arthritis interference in the last month with household work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference).
  The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 321 | 314
units on a scale | 2.7 (2.7) | 2.4 (2.8)

32. Secondary Outcome: Number of Work Days Missed (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of work days missed in the last month. The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Number of work days missed in last month
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 88 | 84
Number of work days missed in last month | 0.2 (0.9) | 0.1 (0.4)

33. Secondary Outcome: Number of Work Days With Reduced Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of work days with reduced productivity in the last month. The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Work days with reduced work productivity
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 88 | 84
Work days with reduced work productivity | 0.6 (2.1) | 0.3 (1.1)

34. Secondary Outcome: Interference With Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: The arthritis interference in the last month with work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference).
  The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 88 | 83
units on a scale | 0.7 (1.4) | 0.5 (1.1)

35. Secondary Outcome: Number of Days With No Household Work (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of days with no household work in the last month. The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days with no household work
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 172 | 180
Days with no household work | 1.1 (3.1) | 1.3 (3.4)

36. Secondary Outcome: Number of Days With Reduced Household Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of days with reduced household work productivity in the last month. The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days with reduced household work
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 172 | 180
Days with reduced household work | 1.3 (3.3) | 1.1 (2.9)

37. Secondary Outcome: Number of Days Missed of Family/Social/Leisure Activities (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of days missed of family/social/leisure activities in the last month. The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Activity days missed
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 172 | 180
Activity days missed | 0.4 (2.5) | 0.2 (0.9)

38. Secondary Outcome: Number of Days With Hired Outside Help (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of days with hired outside help in the last month. The WPS-RA is a 9-item survey measuring the effect of Rheumatoid Arthritis (RA) and its treatment on the patient's work productivity.
Time Frame: Week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days with hired outside help
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 172 | 180
Days with hired outside help | 0.1 (0.6) | 0.3 (2.1)

39. Secondary Outcome: Interference With Household Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: as for outcome 31
Time Frame: Week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Number analyzed (Participants) | 172 | 180
units on a scale | 1.4 (2.0) | 1.2 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from November 2010 through December 2012.
Description: Adverse Event reporting consists of the Safety Set (SS). The Safety Set (SS) consisted of all subjects who received at least 1 dose of study medication.
Arm/Group | RAPID3 to Assess Response to Cimzia | CDAI to Assess Response to Cimzia
Serious Adverse Events (participants affected / at risk) | 32/369 | 39/367
Other Adverse Events (participants affected / at risk) | 126/369 | 115/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAPID3 to Assess Response to Cimzia (N=369) | CDAI to Assess Response to Cimzia (N=367)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 3 (3) | 0 (0)
Spinal pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (4)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Emphysematous cystitis (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Critical illness myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAPID3 to Assess Response to Cimzia (N=369) | CDAI to Assess Response to Cimzia (N=367)
Bronchitis (Infections and infestations) | 10 (10) | 22 (23)
Sinusitis (Infections and infestations) | 28 (34) | 20 (24)
Upper respiratory tract infection (Infections and infestations) | 37 (39) | 38 (41)
Urinary tract infection (Infections and infestations) | 39 (53) | 38 (46)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (33) | 10 (11)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 19 (21) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.